CLINICAL TRIAL: NCT03731299
Title: Are Spatial and Temporal Muscle Synergy Modules Related to Functional Ability After Stroke?
Brief Title: Muscle Synergies After Stroke
Status: Completed | Type: Observational
Sponsor: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Tamaya Van Criekinge, Principal investigator, Universiteit Antwerpen
Other Study IDs: TVC3
Record Dates: First submitted 2018-10-26; First posted 2018-11-06 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Stroke
Keywords: muscle synergies; gait; functional ability
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stroke: Individuals suffered from a haemorrhagic or ischaemic stroke. Diagnosis has to be confirmed on the basis of CT or MRI imaging.
- Healthy adults: Healthy individuals without any neurological or orthopaedic disorder that could influence motor performance and balance

SUMMARY:
The aim of this systematic review was to determine the number of muscle synergies and the distribution of muscle weightings in stroke patients during gait.

DETAILED DESCRIPTION:
The aim of this systematic review was to determine the number of muscle synergies and the distribution of muscle weightings in stroke patients during gait. Although literature has suggested that merging of synergies occurs after stroke and that a larger number of is associated with increased motor function if compared with healthy adults. IIt is still unknown if this hypothesis is also relevant when comparing different functional levels within a stroke population and what functional impact of altered synergies on walking behavior is.

ELIGIBILITY:
Inclusion Criteria Stroke:

1. haemorrhagic or ischaemic stroke diagnosis, confirmed on the basis of CT or MRI imaging;
2. no known history of previous stroke;
3. stroke onset within five months; 4 patients are between 18 and 85 years of age;

Exclusion Criteria Stroke:

1. A score of 20 or higher on the Trunk Impairment Scale which indicates normal truncal function;
2. A score lower than two on the Functional Ambulation Categories (FAC) as patients needed to be able to ambulate without physical support to ensure that gait analysis can be executed safely;
3. Not able to sit independently for 30 seconds on a stable surface;
4. They suffer from other neurological and orthopaedic disorders that could influence motor performance and balance;
5. not able to understand instructions.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Volunteers: community sample Stroke: Rehabilitation Hospital RevArte, primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Amount of muscle synergies derived by non-negative matrix factorization | Once, in the week of inclusion
  Spatial characteristic of muscle synergy compared to healthy adults: the amount of synergies during walking in stroke subjects, the amount of muscles in one synergie and which muscles in one synergy

SECONDARY OUTCOMES:
Distribution of muscle synerigies derived by non-negative matrix factorization | Once, in the week of inclusion
  Temporal characteristic of muscle synergy compared to healthy adults: When are these synergies active during the gait cycle (100%).

CONTACTS AND LOCATIONS:
Overall Officials: Steven Truijen, Prof., Study Director — Universiteit Antwerpen

IPD SHARING:
Plan to Share IPD: No